CLINICAL TRIAL: NCT05227716
Title: Evaluation of the Clinical Response to Magnesium Sulfate as an Adjunct in the Anesthesia
Brief Title: Clinical Response to Magnesium Sulfate as an Adjunct in the Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Lilia Edith Luque Esparza, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R-2021-902-040
Record Dates: First submitted 2021-12-30; First posted 2022-02-07 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia and Analgesia; Magnesium Sulfate
Keywords: Magnesium Sulfate; Anesthesia; Analgesia; Pain, Postoperative; Receptors, N-Methyl-D-Aspartate
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: * Clinical trial: An intervention will be carried out in the population to be studied for the purpose of the research and there will be a control group.
  * Triple blind: Participants and researchers will be unaware of the type of intervention used (administration of MgSO4 or Placebo).
  * Randomized: A list of random numbers will be used to assign patients to study groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind: Participants and researchers will be unaware of the type of intervention used (administration of MgSO4 or Placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulphate (Experimental): Administration of intravenous MgSO4 as an adjunct to anesthesia.
  Dose: 30 mg / kg of MgSO4 IV 15 minutes before induction of anesthesia and 10 mg / kg / h in continuous IV infusion during the operation
  Interventions: Drug: Perioperative magnesium sulfate
- Placebo (Placebo Comparator): Administration of intravenous physiological solution (NaCl 0.9%) as a complement to anesthesia.
  Dose: equivalent to that administered in the MgSO4 group
  Interventions: Drug: Perioperative magnesium sulfate

INTERVENTIONS:
Drug: Perioperative magnesium sulfate — Administration of magnesium sulfate as an adjunct in anesthesia

SUMMARY:
Magnesium sulfate (MgSO4) has multiple desirable effects in an anesthetic procedure, including modulation of the hemodynamic response to surgical stress, perioperative anesthetic and analgesic effect, potentiation of neuromuscular blockade, and central nervous system depression. MgSO4 is an antagonist of the N-methyl-d-aspartic acid (NMDA) receptor, therefore it produces an analgesic effect related to the prevention of central sensitization caused by peripheral tissue damage.

Objective. To evaluate the perioperative clinical response to MgSO4 as an adjunct to anesthesia.

Material and method. Randomized, triple-blind clinical trial that will include men and women over 18 years of age, scheduled for surgery under general or regional anesthesia. After accepting and signing the informed consent, all patients will be subjected to the same pre, trans and postoperative protocol and will be assigned to 2 groups according to the intravenous administration of MgSO4 (placebo and MgSO4). A brief preoperative medical history will be taken, a peripheral blood sample will be taken to determine preoperative serum Mg, the clinical effect of MgSO4 on trans and postoperative analgesia (EVAD), hemodynamic stability (blood pressure (BP) and heart rate ( HR)), motor and neuromuscular block time (Bromage and TOF), and recovery time. The presence of adverse reactions to anesthesia (nausea, vomiting, chills, pruritus, urinary retention, arrhythmias, laryngeal or bronchial spasm) and those secondary to the administration of Mg, SO4, as well as the total doses of all drugs used during the perioperative. The data will be analyzed in the SPSS software.

DETAILED DESCRIPTION:
The participant selection process will be carried out through direct invitation to patients scheduled for surgery under regional or general anesthesia at the General Hospital of Zone No. 51 of the IMSS, Gómez Palacio, Durango. Explaining what their participation consists of for the subsequent signing of the informed consent letter in case of accepting. Afterwards, according to the type of surgery and scheduled anesthesia, 2 groups will be integrated randomly and blindly for the investigator: one that will receive MgSO4 pre and intraoperatively and another group that will be administered 0.9% NaCl intravenously (placebo). All participants will undergo the same pre, trans and postoperative surgical and anesthetic protocol.

Personal data, background and sociodemographic variables will be collected in a data collection sheet. Subsequently, anthropometric measurements will be made to determine weight, height, body mass index and blood pressure.

Peripheral venous blood samples will be taken in the operating room for the determination of pre and postoperative serum Mg and other analyzes.

Each participant will receive standard and continuous monitoring (electrocardiogram, oxygen saturation, blood pressure, capnography, temperature and TOF) and an intravenous access will be established. The MgSO4 group will receive 30 mg / kg of magnesium sulfate intravenously over a period of 15 minutes before induction of anesthesia and 10 mg / kg / h by continuous intravenous infusion during the operation. The control group (placebo) will receive 0.9% NaCl in the same volume as the study drug.

In procedures under general anesthesia, a standard protocol with propofol 2 mg / kg (IV), fentanyl 2 μg / kg (IV) and cisatracurium 0.2 mg / kg (IV) will be applied. Anesthesia will be maintained with 100% oxygen, and 0.5 to 4 vol% sevoflurane, to achieve a mean alveolar concentration (MAC) of 50%. Maintenance doses of fentanyl will be added to the anesthesia regimen as needed. The maintenance dose of cisatracurium will be administered according to the MNM with TOF. The total doses of the drugs used will be recorded. In cases with neuraxial regional anesthesia, a standard protocol with 10 mg heavy bupivacaine and subarachnoid buprenorphine 60 mcg will be applied.

Hemodynamic parameters will be recorded at baseline (before administration of magnesium sulfate or 0.9% isotonic saline solution and subsequently every 5 minutes during surgery, up to 180 minutes after drug administration.

Low blood pressure during surgery, defined as a mean blood pressure value <50 mmHg, will be treated with a 5 mg bolus of ephedrine given intravenously or norepinephrine by IV infusion for persistent hypotension (this is the standard anesthetic management of variations in hemodynamic stability). Low heart rate during surgery, defined as <50 beats per minute, will be treated with atropine at 10 mcg / kg intravenously.

The time until the MNM with TOF indicates the suitability of the neuromuscular block for intubation will be recorded, and the intubation conditions will be evaluated.

The postoperative analgesic protocol will include ketorolac 30mg IV, tramadol 100mg IV, or lysine clonixinate 100mg in case of allergy to ketorolac. Buprenorphine will be administered subcutaneously at a dose of 2 mcg / kg as rescue analgesia only when necessary.

As an adjunct to anesthesia, dexamethasone 8 mg IV, metoclopramide 10 mg IV, ondansetron 100 mcg / kg and omeprazole 40 mg IV will be administered.

Post-operative pain assessment will be performed by EVAD upon exiting anesthesia and at 2, 4, 6, and 24 hours.

The time elapsed until the first request for additional analgesic by the patient, and the total consumption of postoperative analgesics will be recorded, recording it as morphine equivalents.

All the information about all the drugs administered to the patient during their perioperative stay will be collected.

Episodes of nausea, vomiting, itching, chills, arrhythmias, laryngeal or bronchial spasm will be recorded during and after coming out of anesthesia and at the end of the hospital stay.

Satisfaction in recovery from anesthesia will be assessed at 24 hours by delivering a self-report questionnaire to patients.

Finally, the data will be captured in a database for subsequent statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery under general or regional anesthesia at Hospital General de Zona No. 51.
* Physical state ASA 1 and 2
* BMI 18-30 kg / m2
* Acceptance and signing of the informed consent.

Exclusion Criteria:

* Treatment with calcium or magnesium channel blockers
* Drug use or alcoholism referred by the patient in the questioning
* Neurological diseases
* Myopathy
* Intracardiac block
* Renal insufficiency
* Liver failure
* Pregnancy
* Hematological disorders
* Contraindications to the use of magnesium sulfate (hypersensitivity to the active principle or to any of the excipients, concomitant use with quinidine derivatives, tachycardia, heart failure, myocardial injury, infarction).

Elimination criteria:

* Survey with incomplete data corresponding to the study variables.
* Revocation of informed consent or decision to withdraw by of the patient.
* Loss to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in postoperative analgesia over 24 hours | 15 minutes after coming out of anesthesia, 2, 4, 6 and 24 hours after coming out of anesthesia
  Postoperative pain intensity reported by the participant using the visual analog scale after intravenous infusion of magnesium sulfate or placebo (NaCl at 0.9%).
Time to first request for pain reliever | 24 hours after departure from anesthesia
  Time (minutes) to request analgesia after coming out of anesthesia after intravenous infusion of magnesium sulfate or placebo (NaCl at 0.9%).
Hemodynamic stability | 180 minutes intraoperatively
  Changes in heart rate (beats per minute) and mean systemic arterial pressure (mmHg) intraoperatively after or during intravenous infusion of magnesium sulfate or normal saline (0.9% NaCl) were combined to report hemodynamic stability.
  Changes in heart rate (beats per minute) and mean systemic arterial pressure (mmHg) of less than 20% without the need to administer atropine, ephedrine or other positive chronotropic agents and/or vasoactive agents are considered criteria of hemodynamic stability.
Interaction with neuromuscular blockers (BNM): Onset time | 180 minutes intraoperatively
  Parameters measured per train of four after administration of the non-depolarizing muscle relaxant according to the parameters established in the current guidelines for good clinical research practices in pharmacodynamic studies of neuromuscular blocking agents II:
  - Onset time (OT): Time elapsed from the administration of BNM to obtaining a depression in the monitored motor response of between 80 to 100% with the T1 stimulus pattern of TOF.
Interaction with neuromuscular blockers (BNM):Clinical effect time | 180 minutes intraoperatively
  Parameters measured per train of four after administration of the non-depolarizing muscle relaxant according to the parameters established in the current guidelines for good clinical research practices in pharmacodynamic studies of neuromuscular blocking agents II:
  - Clinical effect time: Time elapsed from administration of BNM until 25% is recovered in the monitored motor response measured with TOF as T1> 25% or ST> 25%.
Interaction with neuromuscular blockers (BNM): Recovery index (RI) | 180 minutes intraoperatively
  Parameters measured per train of four after administration of the non-depolarizing muscle relaxant according to the parameters established in the current guidelines for good clinical research practices in pharmacodynamic studies of neuromuscular blocking agents II:
  - Recovery index (RI): Time elapsed between recovery of 25% and 75% of T1 from TOF.
Adverse reactions to magnesium sulfate | From the start of the magnesium sulfate infusion until 24 hours after leaving anesthesia
  Adverse reactions to the perioperative administration of parenteral magnesium sulfate that derive from magnesium poisoning or alterations in the administration site.
  Administration site alterations (injection site pain, hypothermia, vasodilation with a sensation of heat).
  Nervous system (loss of tendon reflex, headache, dizziness, coma, drowsiness and confusion, CNS depression, respiratory paralysis).
  Cardiovascular system (circulatory collapse, arrhythmias, cardiac arrest).
  Respiratory system (respiratory depression secondary to neuromuscular block).
  Gastrointestinal system (nausea and vomiting).
  Musculoskeletal and connective tissue system (muscle weakness).
  Others (problems with speech, vision, excessive sweating, thirst, or others not reported).
Adverse reactions to anesthesia | 180 minutes intraoperatively up to 24 hours after discharge from anesthesia
  Side and adverse effects associated with the use of anesthetic drugs.
  Nausea, vomiting, itching, chills, urinary retention, arrhythmias, laryngeal or bronchial spasm.
Number of participants carrying polymorphisms related to perioperative clinical response to magnesium sulfate | During the 3-year duration of the study
  Determination of polymorphisms related to the pharmacokinetics of opioids (gene CYP3A4/*16, CYP3A4/*1B), the NMDA receptor (GENE NR1/GRIN1, NR2/GRIN2A, NR2B/GRIN2B, NR3A/GRIN3A, NR3B/GRIN3B), and magnesium transporters (gene CNNM2, TRPM6, SLC41A1, SLC41A2).

SECONDARY OUTCOMES:
Conditions for endotracheal intubation | 5 minutes after the administration of BNM
  Evaluation of the conditions for orotracheal intubation. Use a qualitative scoring system. The factors that are taken into consideration are: ease of laryngoscopy, position and / or movement of the vocal cords and reaction to intubation.
Consumption of intraoperative analgesics | 180 minutes intraoperatively
  Consumption of analgesics (μg of fentanyl) intraoperatively in induction and / or maintenance after / during intravenous infusion of magnesium sulfate or placebo (NaCl at 0.9%), in each group of patients.
Postoperative analgesic consumption | From exit from anesthesia up to 24 hours
  Consumption of opioid analgesics (evaluated as mg morphine equivalents) postoperatively after intravenous infusion of magnesium sulfate or placebo (NaCl at 0.9%).
Consumption of neuromuscular relaxant | 180 minutes intraoperatively
  Consumption of neuromuscular relaxant (mg of cisatracurium) intraoperatively in intubation and / or maintenance after / during intravenous infusion of magnesium sulfate or placebo (0.9% NaCl), in each study group.
Hypnotic use | 180 minutes intraoperatively
  Hypnotic consumption (mg of propofol) intraoperatively in intubation and / or maintenance after / during intravenous infusion of magnesium sulfate or placebo (NaCl at 0.9%), in each study group.
Satisfaction in recovery from anesthesia | 24 hours after departure from anesthesia
  The overall satisfaction of the patients was evaluated the day after surgery using the IOWA scale (Dissatisfied: -3-2-1, Satisfied + 1 + 2 + 3) after intravenous infusion of magnesium sulfate or placebo (NaCl at 0.9%).

OTHER OUTCOMES:
Serum magnesium | Before IV infusion of MgS04 or placebo (NaCl at 0.9%) and 24 hours after coming out of anesthesia
  Serum magnesium concentrations(mg / dL)

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Instituto Mexicano Del Seguro Social, Gómez Palacio, Durango
  - Lilia Edith Luque-Esparza, Gómez Palacio, Durango

IPD SHARING:
Plan to Share IPD: Undecided
This item has not yet been defined